CLINICAL TRIAL: NCT00202215
Title: A Study on the Effects of a Personality Disorder Day Hospital Program on Clients Body Mass Index
Brief Title: Chrysalis Day Program Body Mass Index Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDS002
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2005-09

CONDITIONS: Borderline Personality Disorder; Eating Disorders
Keywords: Day hospital treatment
MeSH Terms: conditions — Borderline Personality Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Chrysalis Day Program

SUMMARY:
This is a study to determine if the approach taken to treat patients in the Chrysalis Day Hospital Program will favourably effect their health status as assessed by Body Mass Index (BMI)

DETAILED DESCRIPTION:
As part of the Providence Continuing Care Center's continuing quality improvement initiatives this study is to more systematically evaluate the success of the Chrysalis Day Hospital Program in dealing with some features of eating disorders commonly experienced by its patients.

At intake all clients will be approached to give informed consent to participate. If they do consent they will have their height and weight recorded( if they request they will not be told their weight)as part of the usual intake process conducted by a dietician.

When clients exit the program they again will be approached to be weighed. The body mass index will be calculated and compared to admission values.

The Chrysalis Program is a unique day hospital approach to treating individuals with severe personality disorders (primarily Borderline)that views the eating disordered behaviour common to these clients as a symptom of many and by addressing core issues of affect dysregulation as well as psychoeducation about eating the eating problems will improve .

ELIGIBILITY:
Inclusion Criteria:

* clients of the Chrysalis Program

Exclusion Criteria:

* clients of the Chrysalis Program who do not consent to the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2001-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Body Mass Index at time of enrolling in programme and at leaving | at entry and upon leaving the program

SECONDARY OUTCOMES:
patient demographics relationship to outcome | upon entry and exit from the program
programme changes and relation to outcome | from start to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H McNevin, MD, Principal Investigator — Queens University
Locations (1):
- Providence Care Centre Mental Health Services, Kingston, Ontario, Canada